CLINICAL TRIAL: NCT03129568
Title: A Prospective Phase 1 Trial of Cardiac Progenitor Cell Therapy in Children With Dilated Cardiomyopathy
Brief Title: Transcoronary Infusion of Cardiac Progenitor Cells in Pediatric Dilated Cardiomyopathy
Acronym: TICAP-DCM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Okayama University (Other)
Collaborators: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Responsible Party: Principal Investigator, Hidemasa Oh, MD, Professor, Okayama University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01F1701003
Record Dates: First submitted 2017-04-14; First posted 2017-04-26 (Actual); Results first posted 2021-11-01 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Dilated Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Intervention Model Description: Transcoronary infusion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CDC infusion (Experimental): CDCs infusion by coronary intervention.
  Interventions: Biological: CDC infusion

INTERVENTIONS:
Biological: CDC infusion — Injection of CDCs (0.3 million per kg of body weight).

SUMMARY:
A phase 1 prospective study to determine the procedural feasibility and safety and preliminary efficacy of intracoronary infusion of cardiosphere-derived cells (CDCs) in patients with dilated cardiomyopathy.

DETAILED DESCRIPTION:
Five consecutive patients will be enrolled to a phase 1 study to verify the procedural feasibility and safety with the CDC infusion group.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as dilated cardiomyopathy.
* Patients aged under 18 years old.
* Cardiac ejection fraction < 40%.

Exclusion Criteria:

* Contradiction to cardiac magnetic resonance imaging.
* Cardiogenic shock.
* A patient with unstoppable extracorporeal circulation.
* A patient with lethal, uncontrollable arrhythmia.
* A patient with a complication of coronary artery disease.
* A patient with a complication of brain dysfunction due to circulatory failure.
* A patient with malignant neoplasm.
* A patient with a complication of a serious neurologic disorder.
* A patient with high-grade pulmonary embolism or pulmonary hypertension.
* A patient with high-grade renal failure.
* A patient with multiple organ failure.
* Active infection (including endocarditis).
* Sepsis.
* Active hemorrhagic disease (e.g. gastrointestinal bleeding, injury).

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2020-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Uemura, M.D., Ph.D., Study Chair — Shonan Tobu Clinic
Locations (1):
- Okayama University Hospital, Okayama, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ishigami S, Ohtsuki S, Eitoku T, Ousaka D, Kondo M, Kurita Y, Hirai K, Fukushima Y, Baba K, Goto T, Horio N, Kobayashi J, Kuroko Y, Kotani Y, Arai S, Iwasaki T, Sato S, Kasahara S, Sano S, Oh H. Intracoronary Cardiac Progenitor Cells in Single Ventricle Physiology: The PERSEUS (Cardiac Progenitor Cell Infusion to Treat Univentricular Heart Disease) Randomized Phase 2 Trial. Circ Res. 2017 Mar 31;120(7):1162-1173. doi: 10.1161/CIRCRESAHA.116.310253. Epub 2017 Jan 4. PMID 28052915
- [Background] Tarui S, Ishigami S, Ousaka D, Kasahara S, Ohtsuki S, Sano S, Oh H. Transcoronary infusion of cardiac progenitor cells in hypoplastic left heart syndrome: Three-year follow-up of the Transcoronary Infusion of Cardiac Progenitor Cells in Patients With Single-Ventricle Physiology (TICAP) trial. J Thorac Cardiovasc Surg. 2015 Nov;150(5):1198-1207, 1208.e1-2. doi: 10.1016/j.jtcvs.2015.06.076. Epub 2015 Jul 8. PMID 26232942
- [Background] Ishigami S, Ohtsuki S, Tarui S, Ousaka D, Eitoku T, Kondo M, Okuyama M, Kobayashi J, Baba K, Arai S, Kawabata T, Yoshizumi K, Tateishi A, Kuroko Y, Iwasaki T, Sato S, Kasahara S, Sano S, Oh H. Intracoronary autologous cardiac progenitor cell transfer in patients with hypoplastic left heart syndrome: the TICAP prospective phase 1 controlled trial. Circ Res. 2015 Feb 13;116(4):653-64. doi: 10.1161/CIRCRESAHA.116.304671. Epub 2014 Nov 17. PMID 25403163
- [Result] Hirai K, Ousaka D, Fukushima Y, Kondo M, Eitoku T, Shigemitsu Y, Hara M, Baba K, Iwasaki T, Kasahara S, Ohtsuki S, Oh H. Cardiosphere-derived exosomal microRNAs for myocardial repair in pediatric dilated cardiomyopathy. Sci Transl Med. 2020 Dec 9;12(573):eabb3336. doi: 10.1126/scitranslmed.abb3336. PMID 33298561

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CDC Infusion
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Consecutive enrollment of 5 patients to receive CDC infusion
Arm/Group | CDC Infusion
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.4 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Cardiac Function [Mean (Standard Deviation); unit: percentage of baseline ejection fraction] | 28.5 (10.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Cardiac Adverse Events Related to Transcoronary Infusion of CDCs.
Description: Assessment of major adverse cardiac events include death, sustained/symptomatic ventricular tachycardia, aggravation of heart failure, acute coronary syndrome, unplanned cardiovascular operation for cardiac tamponade and infection in the first month after injection, and serially afterwards.
Time Frame: 6 months after CDC treatment
Population: Adverse events
Measure: Count of Participants; unit: Participants
Arm/Group | CDC Infusion
Number analyzed (Participants) | 5
Participants | 1

2. Secondary Outcome: Change in Ejection Fraction
Description: To determine the changes in cardiac function by ejection fraction with cardiac MRI evaluation in CDC-treated participants from baseline to 6 months of follow up.
Time Frame: 6 months after protocol treatment
Population: Changes in cardiac function
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | CDC Infusion
Number analyzed (Participants) | 5
percentage of ejection fraction | 4.5 (10.2)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | CDC Infusion
All-Cause Mortality (participants affected / at risk) | 1/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CDC Infusion (N=5)
heart failure (Cardiac disorders) | 1 (1)
infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ischemic event (Cardiac disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Single arm study without placebo control comparator

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT03129568/Prot_SAP_000.pdf